CLINICAL TRIAL: NCT00627003
Title: A Double-blind, Randomized, Placebo-controlled Multicenter Efficacy Study for the Treatment of Patients With Restless Legs Syndrome (RLS)
Brief Title: A Study to Evaluate the Efficacy and Safety of Cabergoline Compared With Placebo for the Treatment of RLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CABAS-0067-033
Record Dates: First submitted 2008-02-19; First posted 2008-02-29 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cabergoline
- 2 (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cabergoline — Cabergoline oral tablets administered once daily in the evening: 0.5 mg daily on Days 1 to 3, 1.0 mg daily on Days 4 to 7, 1.5 mg daily on Days 8 to 10, and 2.0 mg daily on Days 11 to 14, followed by a stable dose for an additional 3 weeks
  Arms: 1
Other: Placebo — Placebo oral tablets administered daily for 5 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cabergoline compared with placebo on periodic leg movements (PLMS) arousl index and sleep efficiency in patients with RLS. Also, additional objective and subjective sleep parameters and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic RLS
* Moderate to severe symptoms as indicated by an IRLS total score greater than or equal to 10 and a severity at night score of greater than or equal to 4
* In a baseline polysomnography, patients had to have periodic leg movements during sleep arousal index greater than 5/hour of total sleep time

Exclusion Criteria:

* Patients suffering from seconadry RLS, due to causes such as iron deficiency or renal disease, or suffering from secondary RLS while taking drugs suspected of causing secondary forms of RLS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-11; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | Week 5
PLMS-arousal index (PLMS-AI) | Week 5

SECONDARY OUTCOMES:
Sleep Questionnaire Form A | Weeks 2 and 5
Quality of Life for RLS questionnaire | Weeks 2 and 5
Clinical Global Impressions | Weeks 2 and 5
Safety including type and frequency of adverse events, changes in laboratory data and abnormalities observed in electrocardiography | Weeks 2 and 5
Total score of the severity rating scale of the International RLS (IRLS) Study Group | Weeks 2 and 5
RLS-6 severity scales | Weeks 2 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CABAS-0067-033&StudyName=A%20study%20to%20evaluate%20the%20efficacy%20and%20safety%20of%20cabergoline%20compared%20with%20placebo%20for%20the%20treatment%20of%20RLS%20